CLINICAL TRIAL: NCT00815620
Title: Best Therapy for Patients With Neuroendocrine Tumors
Acronym: BESTTHERAPYNET
Status: Completed | Type: Observational
Sponsor: Zentralklinik Bad Berka (Other)
Responsible Party: Principal Investigator, Dieter Hoersch MD, Senior consultant, Zentralklinik Bad Berka
Other Study IDs: ZBB-NET-1
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumors; transcatheter arterial chemoembolization; selective internal radiotherapy; surgery; radio-frequency ablation; peptide-receptor radiotherapy; progression-free survival; quality of life; overall survival; weight; time of hospitalization
MeSH Terms: conditions — Neuroendocrine Tumors; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: patients undergoing local ablative therapy such as transcatheter-arterial chemoembolization or selective interal radiotherapy
- 2: patients undergoing surgery or radiofrequency ablation
- 3: patients undergoing peptide receptor radiotherapy

SUMMARY:
A prospective observational study containing three arms comprising different therapeutic measures to treat patients with neuroendocrine tumors in advanced stages. The therapy arms include local ablative therapy such as TACE or SIRT, surgery and RFA with peptide receptor radiotherapy.

DETAILED DESCRIPTION:
Study design:

Prospective observational study comparing ablative measures as TACE or SIRT with surgery/RFA and with peptide receptor radio-therapy in patients with advanced well-differentiated neuroendocrine tumors with lymph node or distant metastases (N1, M1) Prospective evaluation Primary end points: time to progression Secondary end points: survival, quality of life (EORTC-QLQ30), weight, time of hospitalization, Karnofsky index) Non-randomized cohort study Number of patients needed in all groups: 70 per group, 210 overall Evaluation of response to therapy every 3-6 months by imaging, clinical status, weight, quality of life, Karnofsky-index Cross-over allowed if therapy changes

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven neuroendocrine tumor (WHO class I-II, TNM grading 1-2)
* Advanced disease with lymph node or distant metastases (N1, M1) undergoing cytoreduction by surgery/local ablative therapy or peptide receptor radiotherapy
* curative intent of all therapies possible

Exclusion Criteria:

* Undifferentiated neuroendocrine carcinoma (WHO class III, TNM grading 3)
* secondary tumor
* advanced carcinoid heart disease requiring surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with neuroendocrine tumors in a tertiary referal center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-11; Primary Completion 2016-08 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 2 years

SECONDARY OUTCOMES:
overall survival, quality of life (EORTC-QLQ30), weight, time of hospitalization, Karnofsky index | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hörsch, MD, Principal Investigator — Zentralklinik Bad Berka GmbH
Locations (1):
- Zentralklinik Bad Berka, Bad Berka, Germany